CLINICAL TRIAL: NCT03801837
Title: Macadamia Nut Effects on Adiposity and Cardiometabolic Risk Factors
Brief Title: Effect of Macadamia Nut on Cardiometabolic Risk Factors
Acronym: MAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, Joan Sabate,DrPH, MD, Professor of Nutrition, Loma Linda University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 5190008
Record Dates: First submitted 2019-01-07; First posted 2019-01-14 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Risk Factor; Heart Diseases; Inflammation
Keywords: Macadamia Nuts; Cardiovascular Disease; Inflammation
MeSH Terms: conditions — Heart Diseases; Inflammation; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Macadamia Nut Diet (Active Comparator): This group will have their habitual diet supplemented with appropriate portion of Macadamia Nuts (15% of daily calories or 30-45 grams based on Kcal requirement of the individual)
  Interventions: Dietary Supplement: Macadamia Nut
- Control Diet (Placebo Comparator): This group will continue with their Habitual Diet
  Interventions: Dietary Supplement: Control Diet

INTERVENTIONS:
Dietary Supplement: Macadamia Nut — Participants will be provided with the appropriate portion of macadamia nuts [15% of daily calories or 30-45 grams based on kcal requirement of the individual]
  Arms: Macadamia Nut Diet
Dietary Supplement: Control Diet — Participants will continue with their Habitual Diet during this part of the intervention
  Arms: Control Diet

SUMMARY:
This research study will test the effects of macadamia nuts on adiposity, and traditional and emergent risk factors of cardiometabolic disease in adult men and women

DETAILED DESCRIPTION:
Purpose of this study is to investigate the effects of Macadamia nuts on body weight, adiposity, , oxidative stress, glucose, insulin an lipid levels. it will a randomized cross over study that will include two study diets (Macadamia nut diet and control diet) with a wash out period of 4 weeks in between. 40 subjects will be selected and randomized into either of the two phases. During the Macadamia nut diet phase subjects will be provided the appropriate portion of Macadamia nuts (15% of daily calories or 30-45 grams based on kcal requirement of the individual, instructions will be provided on how to incorporate nuts into the diet. this phase will last for 8 weeks. During the control diet phase, subjects will continue with their normal diet and abstain from eating nuts. subjects will be tested for various outcomes at baseline and twice at the end of each phase. The intervention will last for 5 months in total.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and post-menopausal women
* Overweight (BMI 25-<40)
* Waist circumference ≥88.9 cm for women and ≥101.6 cm for men
* At least one of the following within the past year:
* Plasma triglycerides ≥150mg/dl
* Blood Pressure ≥130/85 mmHg or participants taking Antihypertensive medication
* Fasting glucose ≥100 mg/dL
* Low Density Lipoproteins>= 130 mg/dl

Exclusion Criteria:

* Nut allergy, any
* Significant chronic disease including: diabetes, congestive heart failure, renal failure, cirrhosis, or autoimmune disease
* Medications affecting lipid or glucose metabolism, immune modulators, or antibiotics in the last 6 months
* Mega-doses of lipid-lowering dietary supplements in the last 6 months
* Cancer in the last 10 years (with the exception on non-melanoma skin cancer)
* Pregnancy or lactation
* Weight change of >10% of body weight in the last 3 months.
* Tobacco use
* Claustrophobia (may affect BOD POD testing)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-11-25 (Actual)

PRIMARY OUTCOMES:
change in body weight | baseline to 18 weeks
  The objective of this measure is to see if eating macadamia nuts could reduce body weight. An In body machine will be used to identify this by measuring the weight of the participants at the baseline and at the end of each diet phase. The weight will be measured in Kilograms
change in body adiposity | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia Nuts could reduce percentage body fat. Air Displacement Plethysmography will be used to determine any change in body percentage fat at the baseline and end of each diet phase
change in body fat mass | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia nuts could change body fat mass at the baseline and end of each diet phase using In Body device (InBody570, Seoul, Korea) that utilizes bioelectric impedance method.
change in body percentage fat | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia nuts could change body percentage fat at the baseline and end of each diet phase using In Body device (InBody570, Seoul, Korea) that utilizes bioelectric impedance method.
change in total body water | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia nuts could change total body water at the baseline and end of each diet phase using In Body device (InBody570, Seoul, Korea) that utilizes bioelectric impedance method.
change in skeletal muscle mass | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia nuts could change skeletal muscle mass at the baseline and end of each diet phase using In Body device (InBody570, Seoul, Korea) that utilizes bioelectric impedance method.
change in lean body mass | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia nuts could change lean body mass at the baseline and end of each diet phase using In Body device (InBody570, Seoul, Korea) that utilizes bioelectric impedance method.
change in dry lean mass | baseline to 18 weeks
  The objective of this measure is to see if eating Macadamia nuts could change dry lean mass at the baseline and end of each diet phase using In Body device (InBody570, Seoul, Korea) that utilizes bioelectric impedance method.
change in fasting plasma cholesterol (mg/dl) | baseline to 18 weeks
  change in fasting plasma cholesterol (mg/dl) will be measured by an enzymatic method with the use of a single aqueous reagent
change in fasting plasma low density lipoprotein cholesterol (mg/dl) | baseline to 18 weeks
  change in fasting plasma low density lipoprotein cholesterol (mg/dl) will be estimated by the use of a two reagent calorimetric enzymatic homogeneous system on the AU480 clinical chemistry analyzer
change in fasting plasma high density lipoprotein cholesterol (mg/dl) | baseline to 18 weeks
  change in fasting plasma high density lipoprotein cholesterol (mg/dl) will be measured by a two-phase reaction with calorimetric end point detection
change in fasting plasma triglycerides(mg/dl) | baseline to 18 weeks
  change in fasting plasma triglycerides(mg/dl) will be measured by an enzymatic hydrolysis method
change in serum apolipoprotein B (mg/dl) | baseline to 18 weeks
  change in serum apolipoprotein B (mg/dl) will be measured by an immuno-turbidimetric procedure using AU480 clinical chemistry analyser
change in serum apolipoprotein A1 (mg/dl) | baseline to 18 weeks
  change in serum apolipoprotein A1 (mg/dl) will be measured by an immuno-turbidimetric procedure using AU480 clinical chemistry analyser
change in serum small density low density lipoprotein cholesterol (mg/dl) | baseline to 18 weeks
  change in serum small density low density lipoprotein cholesterol (mg/dl) will be measured using a two reagent calorimetric enzymatic homogenous system on the AU480 clinical chemistry analyzer.
change in serum oxidized low density lipoprotein (mg/dl) | baseline to 18 weeks
  change in serum oxidized low density lipoprotein (mg/dl) will be measured using a sandwich enzyme-linked immunosorbent assay, Human oxidized low density lipoprotein enzyme linked immunosorbent assay kit
change in fasting plasma glucose | baseline to 18 weeks
  change in fasting plasma glucose levels (mg/dl) will be measured on a clinical chemistry analyzer,AU480 Clinical Chemistry Analyzer, (Beckman Coulter, Inc., Diagnostics Division Headquarters, Brea CA 92821.)
change in fasting plasma insulin | baseline to 18 weeks
  change in fasting plasma insulin (uIU/ml) will be measured measured by solid-phase, two-site chemiluminescent immunometric assays using the IMMULITE 2000, (Siemens Healthcare Diagnostics, Los Angeles, CA 90045)
change in insulin resistance | baseline to 18 weeks
  change in insulin resistance will be measured using the Homeostatic Model Assessment calculator version 2 (HOMA2-IR)

SECONDARY OUTCOMES:
effect modification of adiposity | baseline to 18 weeks
  The objective of this measure is to determine if adiposity is an effect modifier of low density lipoprotein cholesterol, lowering the effect of the macadamia nut intake. The test of this interaction will be performed using statistical analysis system (SAS) software
change in serum Interleukin -6 | baseline to 18 weeks
  change in serum interleukin-6 (pg/ml) will be measured by enzyme linked immunosorbent assay(ELISA)
change in serum tumor necrosis factor alpha | baseline to 18 weeks
  change in serum tumor necrosis factor alpha (pg/ml) will be measured by enzyme linked immunosorbent assay(ELISA)
change in serum soluble selectin (ng/ml) | baseline to 18 weeks
  change in serum soluble selectin (ng/ml) will be measured by enzyme linked immunosorbent assay(ELISA)
change in serum soluble -intercellular adhesion molecule 1 (ng/dl) | baselline to 18 weeks
  change in serum soluble -intercellular adhesion molecule 1 (ng/dl)will be measured by enzyme linked immunosorbent assay(ELISA)
change in serum soluble -vascular adhesion molecule 1 (ng/dl) | baselline to 18 weeks
  change in serum soluble -intercellular adhesion molecule 1 (ng/dl)will be measured by enzyme linked immunosorbent assay(ELISA)
change in C reactive protein | baseline to 18 weeks
  change in C reactive protein (mg/l) will be measured by enzyme linked immunosorbent assay(ELISA)
change in Malondialdehyde | baseline to 18 weeks
  change in Malondialdehyde (micromole/l) will be measured by a competitive enzyme-linked immunosorbent assay
change in Prostaglandin F2 alpha | baseline to 18 weeks
  change in Prostaglandin F2 alpha will be measured by a competitive enzyme-linked immunosorbent assay

CONTACTS AND LOCATIONS:
Overall Officials: Joan Sabate, DrPH, Principal Investigator — Loma Linda University
Locations (1):
- Loma Linda University School of Public Health, Loma Linda, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jones JL, Sabate J, Heskey C, Oda K, Miles F, Rajaram S. Macadamia nut effects on cardiometabolic risk factors: a randomised trial. J Nutr Sci. 2023 May 8;12:e55. doi: 10.1017/jns.2023.39. eCollection 2023. PMID 37180485